CLINICAL TRIAL: NCT05825404
Title: The Effect of Smart Ambient Bright Light for Nursing Home Residents With Alzheimer's Disease and Related Dementias
Brief Title: Smart Lighting for Nursing Home Residents With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Ying-Ling Jao RN, PhD, FGSA, Associate Professor, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00020216
Record Dates: First submitted 2023-03-28; First posted 2023-04-24 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer's Disease and Related Dementias
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: 29 resident participants participated in randomized controlled trial for testing intervention efficacy.
  22 staff participants participated in mixed methods interview for evaluating intervention feasibility.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Smart ambient bright light (Experimental): The smart ambient bright light (SABL) intervention provides auto-controlled, consistent indoor lighting that incorporates natural daylight.
  Interventions: Device: Smart Ambient Bright Light (SABL)
- Control (Sham Comparator): Usual light.
  Interventions: Other: Control

INTERVENTIONS:
Device: Smart Ambient Bright Light (SABL) — The Proposed Smart Ambient Bright Light (SABL) includes tunable LED lights, photosensors, and controllers. The SABL will provide bright light targeted at 400 lux and CS=0.3 in participant bedrooms and designated areas such as the dining room and activity room during the day and provide dim light ≤40 lux and CS≤0.1 in participant bedrooms at night
  Arms: Smart ambient bright light
Other: Control — Usual light.
  Arms: Control

SUMMARY:
This proposed study seeks to develop a smart ambient bright light (SABL) intervention to provide auto-controlled, consistent indoor lighting that incorporates natural daylight. This SABL includes tunable LED lights, photosensors, and controllers. The SABL system has a pre-programmed 24-hour control schedule for illuminance settings to mimic the natural bright-dark cycle. It will automatically adjust the lights to accommodate the daylight effect to minimize staff burden and maximize the LI effect. The SABL will be installed in participants' bedrooms and designated areas in the dining rooms and activity rooms for four weeks. Each participant will wear a personal light monitor to measure the lighting dosage each participant receives. This study will address three aims: 1) pilot test the effect of SABL on reducing agitation in persons with ADRD, 2) evaluate the fidelity of the SABL delivery, and 3) evaluate the feasibility of implementing the SABL. The study will be conducted in two NHs in Pennsylvania. For aims 1 and 2, the investigators will use a crossover, cluster randomized control trial (RCT) and will enroll residents with ADRD and agitation. For aim 3, the investigators will use a mixed methods design and will interview NH stakeholders to evaluate the acceptability, feasibility, and appropriateness of the intervention. This is the first study that incorporates daylight in ambient light interventions and the first study that addresses the measurement, feasibility, and fidelity of lighting interventions. Findings will establish evidence-based implementation strategies and the best design for SABL to reduce agitation for persons with ADRD in NHs.

DETAILED DESCRIPTION:
Up to 90% of people with Alzheimer's disease and related dementias (ADRD) experience at least one behavioral and psychological symptom of dementia (BPSD). Agitation is among the most common and challenging BPSD, especially in nursing home (NH) residents with ADRD. Thus, identifying an effective, non-pharmacological intervention to reduce agitation and other BPSDs is critical. Lighting is important for people with ADRD, especially those living in NHs, as they are not exposed to sufficient daylight. Lighting interventions (LIs) work to regulate suprachiasmatic nuclei, maintain a stable circadian rhythm and reduce agitation. LIs are not invasive and have minimal adverse effects, making them ideal interventions for persons with ADRD. Evidence has reported that LIs show improvement in agitation and other BPSDs for persons with ADRD. However, LIs have not been widely implemented in "real world" care settings. Traditional methods using light boxes that required persons with ADRD to sit and keep their eyes oriented toward a bright light led to compliance and workload issues. A more efficient approach to delivering LIs is necessary. Interest has arisen in designing NHs with the capability of providing LIs via ambient LIs. While a few studies have reported positive effects of ambient LIs on agitation, these studies were conducted in settings with window shades closed to minimize daylight. To establish ambient lighting as a feasible and effective intervention, a few fundamental gaps need to be addressed: 1) a feasible implementation approach to ambient LIs, and 2) intervention fidelity (ensuring the lighting received by participants meets the targets). This proposed study seeks to develop a smart ambient bright light (SABL) intervention to provide auto-controlled, consistent indoor lighting that incorporates natural daylight. This SABL includes tunable LED lights, photosensors, and controllers. The SABL system has a pre-programmed 24-hour control schedule for illuminance settings to mimic the natural bright-dark cycle. It will automatically adjust the lights to accommodate the daylight effect to minimize staff burden and maximize the LI effect. The SABL will be installed in participants' bedrooms and designated areas in the dining rooms and activity rooms for four weeks. Each participant will wear a personal light monitor to measure the lighting dosage each participant receives. This study will address three aims: 1) pilot test the effect of SABL on reducing agitation in persons with ADRD, 2) evaluate the fidelity of the SABL delivery, and 3) evaluate the feasibility of implementing the SABL. The study will be conducted in two NHs in Pennsylvania. For aims 1 and 2, the investigators will use a crossover, cluster randomized control trial (RCT) and will enroll residents with ADRD and agitation. For aim 3, the investigators will use a mixed methods design and will interview NH stakeholders to evaluate the acceptability, feasibility, and appropriateness of the intervention. This is the first study that incorporates daylight in ambient light interventions and the first study that addresses the measurement, feasibility, and fidelity of lighting interventions. Findings will establish evidence-based implementation strategies and the best design for SABL to reduce agitation for persons with ADRD in NHs.

ELIGIBILITY:
Resident participants

Inclusion Criteria:

* Age≥55
* English speaking
* Nursing home residency≥3 months
* Clinical Diagnosis of Alzheimer's Disease and related dementia
* Presence of agitation over the past week

Exclusion Criteria:

* Major sleep problems
* Major mental illness
* Severe vision impairment
* Severe acute or terminal illness

Staff participants:

Inclusion criteria:

* Age≥18
* English speaking
* Employed as a certified nurse assistant (CNA), activity staff, nurse, director of nursing (DON), director of maintenance, administer or other leadership position for at least 3 months. The CNA, activity staff, and nurse must have direct care interactions with the resident participant(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Ling Jao, PhD, Principal Investigator — Penn State University
Locations (2):
- United States (2):
  - Valley View Retirement Community, Belleville, Pennsylvania
  - Christ the King Manor, DuBois, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Figueiro MG, Plitnick B, Roohan C, Sahin L, Kalsher M, Rea MS. Effects of a Tailored Lighting Intervention on Sleep Quality, Rest-Activity, Mood, and Behavior in Older Adults With Alzheimer Disease and Related Dementias: A Randomized Clinical Trial. J Clin Sleep Med. 2019 Dec 15;15(12):1757-1767. doi: 10.5664/jcsm.8078. Epub 2019 Nov 8. PMID 31855161
- [Background] Figueiro MG, Hunter CM, Higgins P, Hornick T, Jones GE, Plitnick B, Brons J, Rea MS. Tailored Lighting Intervention for Persons with Dementia and Caregivers Living at Home. Sleep Health. 2015 Dec 1;1(4):322-330. doi: 10.1016/j.sleh.2015.09.003. PMID 27066526
- [Background] Jao YL, Wang J, Liao YJ, Parajuli J, Berish D, Boltz M, Van Haitsma K, Wang N, McNally L, Calkins M. Effect of Ambient Bright Light on Behavioral and Psychological Symptoms in People With Dementia: A Systematic Review. Innov Aging. 2022 Mar 24;6(3):igac018. doi: 10.1093/geroni/igac018. eCollection 2022. PMID 35602310

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a clustered cross-over RCT design; all participants will be in the intervention and control groups. The study period is 13 weeks, and the sequences were randomly assigned as follows:
  Nursing Home A: Baseline (week 1), SABL (weeks 2-5), post-SABL/washout (weeks 6-7), control/usual light (weeks 8-11), and post control (weeks 12-13).
  Nursing Home B: Baseline (week 1), control/usual light (weeks 2-5), post-control/washout (weeks 6-7), SABL (weeks 8-11), and post intervention (weeks 12-13).
Units Other Than Participants: Nursing home facility
Groups:
- Smart Ambient Bright Light, Then Usual Light: The residents received Smart Ambient Bright Light (weeks 2-5) followed by Usual Light (weeks 8-11) with two weeks of washout period in between (weeks 6-7).
  This is a cluster cross-over RCT design. Two participating nursing homes will be randomly assigned to two study sequences (one site will begin with the intervention period first followed by the control period while the other site will begin with the control period followed by the intervention period). All sites and all participants will be invited to the intervention and control group
  The smart ambient bright light (SABL) intervention provides auto-controlled, consistent indoor lighting incorporating natural daylight.
  Smart Ambient Bright Light (SABL): The Proposed Smart Ambient Bright Light (SABL) includes tunable LED lights, photosensors, and controllers. The SABL will provide bright light targeted at 400 lux and CS=0.3 in participant bedrooms and designated areas such as the dining room and activity room during the day and provide dim light ≤40 lux and CS≤0.1 in participant bedrooms at night.
  Control: usual light
- Usual Light, Then Smart Ambient Bright Light: The residents received usual light first (weeks 2-5) followed by Smart Ambient Bright Light (weeks 8-11) with two weeks of washout period in between (weeks 6-7).
Period: Baseline (Week 1)
Arm/Group | Smart Ambient Bright Light, Then Usual Light | Usual Light, Then Smart Ambient Bright Light
Started | 16; 1 Nursing home facility | 13; 1 Nursing home facility
Completed | 16; 1 Nursing home facility | 13; 1 Nursing home facility
Not Completed | 0; 0 Nursing home facility | 0; 0 Nursing home facility
Period: First Intervention (Weeks 2-5)
Arm/Group | Smart Ambient Bright Light, Then Usual Light | Usual Light, Then Smart Ambient Bright Light
Started | 16; 1 Nursing home facility | 13; 1 Nursing home facility
Completed | 16; 0 Nursing home facility | 12; 1 Nursing home facility
Not Completed | 0; 1 Nursing home facility | 1; 0 Nursing home facility
Not completed — Death | 0 | 1
Period: Washout (Weeks 6-7)
Arm/Group | Smart Ambient Bright Light, Then Usual Light | Usual Light, Then Smart Ambient Bright Light
Started | 16; 1 Nursing home facility | 12; 1 Nursing home facility
Completed | 16; 1 Nursing home facility | 12; 1 Nursing home facility
Not Completed | 0; 0 Nursing home facility | 0; 0 Nursing home facility
Period: Second Intervention (Weeks 8-11)
Arm/Group | Smart Ambient Bright Light, Then Usual Light | Usual Light, Then Smart Ambient Bright Light
Started | 16; 1 Nursing home facility | 12; 1 Nursing home facility
Completed | 16; 1 Nursing home facility | 11; 1 Nursing home facility
Not Completed | 0; 0 Nursing home facility | 1; 0 Nursing home facility
Not completed — Death | 0 | 1
Period: Follow up (Weeks 12-13)
Arm/Group | Smart Ambient Bright Light, Then Usual Light | Usual Light, Then Smart Ambient Bright Light
Started | 16; 1 Nursing home facility | 11; 1 Nursing home facility
Intervention Feasibility, Acceptability, and Appropriateness From Stakeholder Perspectives | 11; 1 Nursing home facility | 11; 1 Nursing home facility
Completed | 16; 1 Nursing home facility | 11; 1 Nursing home facility
Not Completed | 0; 0 Nursing home facility | 0; 0 Nursing home facility

BASELINE CHARACTERISTICS:
Groups:
- Resident Participants: This is a cross-over RCT. All participants are invited to participate in the intervention and control.
  The smart ambient bright light (SABL) intervention provides auto-controlled, consistent indoor lighting that incorporates natural daylight.
  Smart Ambient Bright Light (SABL): The Proposed Smart Ambient Bright Light (SABL) includes tunable LED lights, photosensors, and controllers. The SABL will provide bright light targeted at 400 lux and CS=0.3 in participant bedrooms and designated areas such as the dining room and activity room during the day and provide dim light ≤40 lux and CS≤0.1 in participant bedrooms at night
  Usual light This is a cross-over RCT. All participants will participate in the intervention and control.
- Stakeholder/Staff Participants: At the end of the intervention, we enrolled nursing home stakeholders, including certified nursing assistants, activity staff, nurses, directors of nursing, maintenance, and administrators. 22 participants (11 from each NH)
- Total: Total of all reporting groups
Arm/Group | Resident Participants | Stakeholder/Staff Participants | Total
Number analyzed (Participants) | 27 | 22 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 87.4 (7.5) | 44.5 (10.3) | 68.1 (23.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 27 | 21 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 22 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Lux During Intervention and Control Periods at the Facility Level
Description: Average Lux during Intervention and Control Periods at the facility level This is a cluster crossover RCT design. Two nursing homes were randomly assigned to two different sequences; one nursing home began with the intervention light (weeks 2-5), followed by the control condition (8-11), while the other nursing home began with the control condition (weeks 2-5), followed by the intervention light (week 8-11).
  Data were collected in weeks 1, 3, 5, 7, 9, 11, and 13. Results were combined and categorized as intervention and control periods.
  For the intervention period, the data reported were the average of weeks 3 and 5 for the intervention first group and weeks 9 and 11 for the control first group.
  For the control period, the data reported were the average of weeks 9 and 11 for the intervention first group and weeks 3 and 5 for the control first group.
Time Frame: Intervention: the average of weeks 3 and 5 for the intervention first group and weeks 9 and 11 for the control first group. Control: the average of weeks 9 and 11 for the intervention first group and weeks 3 and 5 for the control first group.
Measure: Mean (Standard Deviation); unit: Lux
Units Other Than Participants: Nursing Home Site
Groups:
- Intervention: Smart Ambient Bright Light: All residents received the Smart Ambient Bright Light (Intervention) either (weeks 2-5) or (weeks 8-11).
- Control: Usual Light: All residents received the Usual Light either during weeks 2-5 or weeks 8-11.
Arm/Group | Intervention: Smart Ambient Bright Light | Control: Usual Light
Number analyzed (Participants) | 27 | 27
Number analyzed (Nursing Home Site) | 2 | 2
Lux | 394.2 (49.70) | 97.4 (23.82)

2. Primary Outcome: Average Circadian Stimulation (CS) Level During Intervention and Control Periods at the Facility Level
Description: Light CS level at the facility level was measured manually on-site.
  This is a cluster crossover RCT design. Two nursing homes were randomly assigned to two different sequences; one nursing home began with the intervention light (weeks 2-5), followed by the control condition (8-11), while the other nursing home began with the control condition (weeks 2-5), followed by the intervention light (week 8-11).
  Data were collected in weeks 1, 3, 5, 7, 9, 11, and 13. Results were combined and categorized as intervention and control periods.
  For the intervention period, the data reported were the average of weeks 3 and 5 for the intervention first group and weeks 9 and 11 for the control first group.
  For the control period, the data reported were the average of weeks 9 and 11 for the intervention first group and weeks 3 and 5 for the control first group.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: CS
Units Other Than Participants: Nursing home site
Groups:
- Intervention: Smart Ambient Bright Light (SABL)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 27
Number analyzed (Nursing home site) | 2 | 2
CS | 0.302 (0.07) | 0.097 (0.02)

3. Primary Outcome: Average Lux During Intervention and Control Periods at the Individual Level
Description: Light level (lux) at the individual level will be measured using a personal light monitor.
  This is a cluster crossover RCT design. Two nursing homes were randomly assigned to two different sequences; one nursing home began with the intervention light (weeks 2-5), followed by the control condition (8-11), while the other nursing home began with the control condition (weeks 2-5), followed by the intervention light (week 8-11).
  Data were collected in weeks 1, 3, 5, 7, 9, 11, and 13. Results were combined and categorized as intervention and control periods.
  For the intervention period, the data reported were the average of weeks 3 and 5 for the intervention first group and weeks 9 and 11 for the control first group.
  For the control period, the data reported were the average of weeks 9 and 11 for the intervention first group and weeks 3 and 5 for the control first group.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lux
Units Other Than Participants: Nursing Home Site
Groups:
- Intervention: Intervention period.
- Control: Control period
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 27
Number analyzed (Nursing Home Site) | 2 | 2
Lux | 406.89 (102.35) | 286.69 (83.50)

4. Primary Outcome: Average Circadian Stimulation (CS) Level During Intervention and Control Periods at the Individual Level
Description: This is a cluster crossover RCT design. Two nursing homes were randomly assigned to two different sequences; one nursing home began with the intervention light (weeks 2-5), followed by the control condition (8-11), while the other nursing home began with the control condition (weeks 2-5), followed by the intervention light (week 8-11).
  Data were collected in weeks 1, 3, 5, 7, 9, 11, and 13. Results were combined and categorized as intervention and control periods.
  For the intervention period, the data reported were the average of weeks 3 and 5 for the intervention first group and weeks 9 and 11 for the control first group.
  For the control period, the data reported were the average of weeks 9 and 11 for the intervention first group and weeks 3 and 5 for the control first group.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: CS
Units Other Than Participants: Nursing Home Site
Groups:
- Intervention: SABL intervention period
- Control: Usual Light Period.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 27
Number analyzed (Nursing Home Site) | 2 | 2
CS | 0.36 (0.09) | 0.24 (0.08)

5. Primary Outcome: Change in Agitation During the Intervention and Control Periods
Description: Agitation was measured using Cohen-Mansfield Agitation Inventory (CMAI) in weeks 1, 3, 5, 7, 9, 11, 13. Total scores range from 29-203; higher scores, more agitation.
  For the intervention, data were the difference between week 1 (pre-intervention) and week 5 (during intervention) for the intervention first group, and data were the difference between weeks 7 (pre-intervention) and week 11 (during intervention) for the control first group.
  For the control, data were the difference between week 7 (pre-control) and week 11 (during control) for the intervention first group, and data were the difference between week 1 (pre-intervention) and week 5 (during intervention) for the control first group.
Time Frame: Intervention: Intervention first group: difference of weeks 1 & 5; Control first group: difference of weeks 7 & 11 Control: Intervention first group: difference of weeks 7 & 11; Control first group: difference of weeks 1 & 5
Measure: Mean (Standard Deviation); unit: Score on the scale
Units Other Than Participants: Nursing Home Site
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 27
Number analyzed (Nursing Home Site) | 2 | 2
Score on the scale | -4.78 (13.55) | -1.48 (13.05)

6. Primary Outcome: Intervention Acceptability
Description: The intervention acceptability of the lighting intervention were measured based on nursing home stakeholders' perspectives using the Acceptability of Intervention Measure (AIM) and followed up by qualitative interviews. The score ranges from 1-5; a higher score indicates a higher level of acceptability.
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Smart Ambient Bright Light: This is a cross-over RCT. All participants are invited to participate in the intervention and control groups.
  The smart ambient bright light (SABL) intervention provides auto-controlled, consistent indoor lighting that incorporates natural daylight.
  Smart Ambient Bright Light (SABL): The Proposed Smart Ambient Bright Light (SABL) includes tunable LED lights, photosensors, and controllers. The SABL will provide bright light targeted at 400 lux and CS=0.3 in participant bedrooms and designated areas such as the dining room and activity room during the day and provide dim light ≤40 lux and CS≤0.1 in participant bedrooms at night.
  Control: Usual light
Arm/Group | Smart Ambient Bright Light
Number analyzed (Participants) | 22
score on a scale | 4.10 (0.93)

7. Primary Outcome: Intervention Feasibility
Description: The intervention feasibility of the lighting intervention will be measured based on nursing home stakeholders' perspectives using the Feasibility of Intervention Measure (FIM) and followed up by qualitative interviews. The total score ranges from 1-5; a higher score indicates a higher level of feasibility.
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smart Ambient Bright Light
Number analyzed (Participants) | 22
score on a scale | 4.40 (0.51)

8. Primary Outcome: Intervention Appropriateness
Description: The appropriateness of the lighting intervention will be measured based on nursing home stakeholders' perspectives using the Intervention Appropriateness Measure (IAM) and followed up by qualitative interviews. The total score ranges from 1-5; a higher score indicates a higher level of appropriateness.
Time Frame: Week 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smart Ambient Bright Light
Number analyzed (Participants) | 22
score on a scale | 3.99 (0.74)

9. Secondary Outcome: Behavioral and Psychological Symptoms of Dementia (BPSD)
Description: BPSD were measured via the Neuropsychiatry Inventory, including delusions, hallucinations, dysphoria, euphoria, anxiety, agitation, apathy, irritability, disinhibition, aberrant motor behaviors, sleep, and appetite. Each symptom score ranges from 0-12, higher scores more severe.
  Data were collected in weeks 1, 3, 5, 7, 9, 11, and 13 Intervention: the difference between weeks 1 (pre-intervention) and 5 (during intervention) for the intervention first group, and the difference between weeks 7 (pre-intervention) and 11 (during intervention) for the control first group.
  Control: the difference between weeks 7 (pre-control) and week 11 (during control) for the intervention first group, and the difference between weeks 1 (pre-control) and 5 (during control) for the control first group.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Nursing Home Site
Groups:
- Intervention: Smart Ambient Bright Light
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 27
Number analyzed (Nursing Home Site) | 2 | 2
units on a scale
  Agitation | -1.11 (3.88) | -0.07 (3.44)
  Anxiety | -1.15 (3.42) | 0.30 (3.77)
  Apathy | -1.04 (3.41) | 0.07 (2.83)
  Appetite | -1.70 (3.54) | 0.63 (1.98)
  Delusion | -1.70 (4.72) | 0.48 (3.79)
  Depression | -1.59 (4.43) | 0.15 (2.33)
  Disinhibition | -1.74 (3.57) | -0.52 (2.62)
  Elation | -0.52 (2.71) | -0.52 (1.53)
  Hallucinations | -1.15 (3.24) | 0.19 (1.73)
  Irritability | -0.48 (3.92) | -0.30 (3.07)
  Motor behaviors | -0.78 (3.15) | -1.11 (4.36)
  Sleep | -2.04 (3.37) | 0.74 (3.50)

10. Secondary Outcome: Affect
Description: Six affects were measured: contentment, interest, pleasure, anxiety/fear, anger, and sadness, using the Philadelphia Geriatric Center Affect Rating Scale. Each affect score ranges from 1 to 5; higher scores, higher levels.
  Two nursing homes were randomly assigned to different sequences; one nursing home began with intervention (weeks 2-5), followed by control (weeks 8-11), while the other nursing home began with control (weeks 2-5), followed by intervention (weeks 8-11).
  Data were collected in weeks 1, 3, 5, 7, 9, 11, and 13. Intervention: the difference between weeks 1 (pre-intervention) and 5 (during intervention) for the intervention first group, and the difference between weeks 7 (pre-intervention) and 11 (during intervention) for the control first group.
  Control: the difference between weeks 7 (pre-control) and 11 (during control) for the intervention first group, and the difference between weeks 1 (pre-intervention) and 5 (during intervention) for the control first group.
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Nursing Home Site
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 27
Number analyzed (Nursing Home Site) | 2 | 2
score on a scale
  Contentment | 0.22 (1.09) | 0.56 (1.09)
  Interest | 0.26 (1.20) | 0.48 (1.09)
  Pleasure | 0.15 (1.20) | 0.44 (1.15)
  Anger | 0 (0.88) | 0.19 (1.08)
  Fear | 0.04 (1.22) | -0.15 (1.32)
  Sadness | -0.19 (1.14) | 0.00 (1.07)

11. Secondary Outcome: Adverse Effects.
Description: Data on intervention-related adverse effects will be collected via inputs from certified nurse assistants (CNAs) using a checklist, which includes deteriorated BPSDs, skin rash, eye irritation, dizziness, nausea, or any other reactions. Each item will be checked as yes or no. Data were collected at weeks 1, 3, 5, 7, 9, 11, and 13. Data across all weeks was combined.
Time Frame: Weeks 1-13 combined
Measure: Number; unit: participants
Units Other Than Participants: Nursing Home Site
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 27
Number analyzed (Nursing Home Site) | 2 | 2
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Weeks 1, 3, 5, 7, 9, 11, 13
Groups:
- Smart Ambient Bright Light: This is a cluster crossover RCT design. Two nursing homes will be randomly assigned into two different sequences; one site will begin with the intervention period, followed by the control period, while the other site will begin with the control period, followed by the intervention period.
  Intervention: Smart Ambient Bright Light (SABL)
- Usual Light: Control: Usual light
Arm/Group | Smart Ambient Bright Light | Usual Light
All-Cause Mortality (participants affected / at risk) | 1/29 | 1/29
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/29
Other Adverse Events (participants affected / at risk) | 3/29 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smart Ambient Bright Light (N=29) | Usual Light (N=29)
Death (Nervous system disorders) | 1 (1) | 1 (1) — Death due to health conditions deterioration.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Smart Ambient Bright Light (N=29) | Usual Light (N=29)
Nausea (General disorders) | 1 | 0 — Medication-related nausea. Not related to the intervention
Pneumonia (General disorders) | 1 | 0
Urinary tract infection (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT05825404/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT05825404/SAP_003.pdf
  • Informed Consent Form (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT05825404/ICF_002.pdf